CLINICAL TRIAL: NCT02687464
Title: A Multicentre, Randomized Controlled Trial Comparing Appendectomy Versus Non-Operative Treatment For Acute Non-Perforated Appendicitis in Children
Brief Title: Appendectomy Versus Non-Operative Treatment For Acute Non-Perforated Appendicitis in Children
Acronym: APPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); Alberta Children's Hospital (Other); Children's Hospital of Western Ontario (Other); St. Justine's Hospital (Other); Children's Hospital of Winnipeg (Unknown); Le Bonheur Children's Hospital (Other); Karolinska University Hospital (Other); Hospital for Children and Adolescents, Finland (Other); University of Southampton (Other); UCL Institute of Child Health (Unknown); KK Women's and Children's Hospital (Other Government); Uppsala University Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Shawn St. Peter, Shawn St. Peter, MD, Director of Research, Department of Surgery, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15100493
Record Dates: First submitted 2016-01-13; First posted 2016-02-22 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Appendicitis
Keywords: Pediatric Surgery; Pediatrics; Randomized controlled trial,; Antibiotics; Cost effectiveness
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-operative treatment group (Experimental): IV fluids, minimum 12 hrs IV antibiotics, minimum 12 hrs clear PO fluids only, regular clinical review. Discharge within 24 hrs after randomization, if study criteria met. If stable but not adequate improvement for discharge, non-operative management continues. If not improved by 48 hrs, appendectomy will be done. Discharge home once vital signs are within normal limits, light oral diet tolerated, adequate oral pain relief and mobile. Total 10 days of antibiotics (IV and oral) following randomization will be given. Antibiotics used vary between centers and will be current standard of care in that center; improving study feasibility and increased generalization of results.
  Interventions: Other: Non-operative treatment
- Appendectomy group (Active Comparator): Laproscopic appendectomy within 18 hrs of randomization. IV antibiotics given from time of randomization and continued post-operatively per the standardized treatment regimen: children with visibly normal appendix or non-perforated acute appendicitis will receive no further antibiotics; children with perforated appendicitis will continue IV antibiotics for a minimum of 3 days and then per local practice. The type of antibiotics used in each center will be identical to those used in the non-operative treatment group.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Other: Non-operative treatment — will receive a minimum of 12 hours intravenous antibiotics and then receive oral antibiotics once they have shown clinical improvement (a total course of 10 days of antibiotics (intravenous and oral). They will be discharged home once they meet a standardized set of criteria to be used in all centers.
  The choice of antibiotics will vary between centers and will be the antibiotic regimen that is current standard of care in that center allowing each center to maintain current protocols will improve study feasibility and increase generalization of the results.
  Arms: Non-operative treatment group
Procedure: Appendectomy — will undergo laparoscopic appendectomy within 18 hours of randomization and will receive intravenous antibiotics per each site's standard care, from the time of randomization and post-operatively according to a defined and standardized treatment regimen based on consensus for this trial.
  Children with a visibly normal appendix or non-perforated acute appendicitis will receive no further antibiotics; children with perforated appendicitis will continue to receive intravenous antibiotics for a minimum of 3 days, and then per local practice. The type of antibiotics used in each center will be identical to those used in the non-operative treatment group and are not specified by the study.
  Other Names: Laparoscopic appendectomy
  Arms: Appendectomy group

SUMMARY:
Rationale and Aim: The standard treatment for acute appendicitis in children is appendectomy. An increasing body of evidence from the adult literature suggests that acute appendicitis may be treated effectively with antibiotics alone, avoiding the need for surgery. The aim of this study is to investigate the effectiveness of non-operative treatment of acute appendicitis in children.

Study design: Pragmatic, parallel-group, unmasked, non-inferiority multicentre randomized controlled trial (RCT).

Patient allocation: Children will be randomly allocated (age 5-16 years) with a diagnosis of acute appendicitis to either laparoscopic appendectomy or treatment with antibiotics. Randomization will be performed using stratification to ensure equal distribution between groups of presenting clinical and demographic features that may influence outcome including gender, duration of symptoms and center.

Interventions: One group of children will undergo laparoscopic appendectomy that is the current standard treatment for children with acute appendicitis. The other group will be treated with intravenous antibiotics. A treatment pathway specifically designed for this study will be used.

Primary Outcome: To be meaningful to parents of, and clinicians treating, children with acute appendicitis, the primary outcome is treatment failure defined as: (i) any additional intervention related to appendicitis requiring general anesthesia within 1 year of randomization (including recurrence of appendicitis after non-operative treatment, which we will treat with appendectomy) or (ii) negative appendectomy. Secondary outcomes are: (i) complications; (ii) time to discharge following randomization; (iii) number and duration of hospital admissions.

Sample size and data analysis: The proposed RCT has a 20% non-inferiority margin to test the null hypothesis that treatment with antibiotics is inferior to appendectomy. Based on data from collaborating centers and a pilot study that we have performed, we expect recruitment of 978 children in total (90% power) over 19 months allowing for drop out. Follow-up will be for 12 months.

DETAILED DESCRIPTION:
Background Acute appendicitis is the commonest surgical emergency in children. The lifetime risk of developing appendicitis is 7-8%, with a peak incidence in the teenage years.The associated financial burden of treating appendicitis is very large.

For over 100 years, surgical removal of the appendix has been deemed necessary to effectively treat acute appendicitis. Appendectomy remains the cornerstone of treatment for acute appendicitis, with the exception of phlegmon or appendix mass. However, in recent years this surgical dogma has been challenged and there is a growing literature to suggest that antibiotics without surgery may be an effective treatment for acute appendicitis in adults and more recently in children. However this non-operative management of acute appendicitis remains controversial and unproven due to the lack of large prospective randomized controlled trials.

Although appendectomy is generally a simple procedure, it requires general anesthesia and is an abdominal operation with inherent risks and potential complications. Complications related to surgery or anesthesia events occur in over 10% of children within 30 days of appendectomy. Although a non-operative approach may avoid these risks and reduce complication rate, this would not be a viable alternative to surgery unless it is equally effective at curing acute appendicitis.

The existing literature relating to the efficacy of non-operative treatment of acute appendicitis in predominantly from adult patients. Several trials and systematic reviews have been reported. A most recent meta-analysis concluded that there were benefits to non-operative treatment including fewer complications, better pain control, and shorter sick leave but that the combined failure and recurrence rate in patients treated non-operatively made this approach less effective overall.

In children, the literature is limited. The most significant studies are: Abes et al [6] who described successful, non-operative treatment in 15 of 16 children who had a very short duration of illness, and minimal diagnostic criteria on imaging; Armstrong et al [7] who reported a 75% success rate in 12 children treated non-operatively along with a matched comparison group undergoing surgery; two RCTs from the USA that compared appendectomy with antibiotic treatment for children with perforated appendicitis [8,9] (a different patient group from the one which we intend to study); a single centre, preference-based, non-randomized study comparing laparoscopic appendectomy with antibiotic treatment [10] that reported interim results only.

In preparation for this multi center RCT, investigators have performed a pilot RCT at one of the participating centers (Karolinska Institute, Stockholm) [11]. Successfully demonstrated feasibility of recruitment to a RCT and safety of non-operative treatment of children with acute appendicitis.

Based on these observations, and in response to parents who are now asking whether their child with acute appendicitis really needs an operation, this randomized controlled trial comparing appendectomy with non-operative treatment in children with acute appendicitis will be done. The principal research question is: Can children with acute uncomplicated (non-perforated) appendicitis be treated without appendectomy?

Rationale for the Trial This trial has the potential to significantly alter clinical practice for one of the most common acute health conditions in children. A finding of non-inferiority of treatment with antibiotics compared to appendectomy would be transformative for the healthcare of children with acute appendicitis in Canada and abroad, including low- and middle-income countries. Reducing the need for surgery in the treatment of childhood appendicitis represents the potential for cost savings for the healthcare system, and will enable improved access for children with non-emergent conditions who are awaiting surgery.

Methods/Design Research question Can children with acute non-perforated appendicitis be treated with antibiotics, rather than appendectomy?

Trial design The APPY trial has been designed as a pragmatic, parallel-group, unmasked, non-inferiority multicentre, international randomized controlled trial. The protocol has been developed in accordance with the SPIRIT guideline and the trial will be conducted and reported according to the CONSORT statement.

Participants Children (5-16 years of age) with suspected acute uncomplicated appendicitis will be enrolled from up to 16 hospitals across Europe and North America. All centers are specialist Pediatric Surgery Referral Centers with trained Specialist Pediatric Surgeons and Pediatric Surgery Training Programs. All children with suspected acute non-perforated appendicitis will be assessed by the on-call surgeon who will determine eligibility for the study. This will be based on a clinical and/or ultrasound diagnosis of acute non-perforated appendicitis. The patient and child will be informed of the trial and invited to participate.

Randomization After signed informed consent, a standardized data set will be collected from all participants at all participating institutions. Patients enrolled in the study will be randomized to groups (1:1 ratio) using an online stratified randomization tool, allowing instant assignment to treatment group 24 hours per day with concealment of allocation. Allocation to groups will be stratified taking into account factors that may affect outcome of treatment: 1) Sex: Male; Female; 2) Duration of symptoms <48hrs; >48hrs; and 3) Center.

Interventions Patients will be allocated to non-operative antibiotic treatment or appendectomy.

Non-operative treatment group: Participants allocated to non-operative treatment will be treated according to a treatment pathway standardized across all centers comprising intravenous fluid treatment, a minimum of 12 hours of intravenous antibiotics, a minimum period of 12 hours taking clear fluid only, and regular clinical review.

During the next clinical rounds, or alternatively approximately 12 hours after randomization, a review of clinical symptoms will be conducted to detect symptoms and signs of significant clinical deterioration including, but not limited to, increased fever, increased tachycardia, and increased pain or tenderness. If the patient is doing well, they may be advanced to regular diet and be assessed for discharge during the same work day, depending on their clinical progression. If they are stable without deterioration but not improved to the point of discharge they will continue with non-operative management. A patient who has not improved after 48 hours of non-operative management will undergo appendectomy. All decisions will be made by the treating physicians and care team with consideration of the input of parents and child where appropriate.

Children in whom non-operative treatment is successful will receive a minimum of 12 hours intravenous antibiotics and then be switched to oral antibiotics once they have shown clinical improvement. They will be discharged home once they meet a standardized set of criteria to be used in all centers: vital signs (including temperature) within normal limits, tolerating a light diet orally, adequate oral pain relief and mobile. They will receive a total course of 10 days of antibiotics (intravenous and oral) following randomization.

Children within the non-operative treatment group will remain under the care of an attending pediatric surgeon who retains overall responsibility for their care. If a child's clinical condition deteriorates at any time, they will undergo laparoscopic appendectomy, and will receive post-operative care identical to that of children in the appendectomy treatment group (see below), and any other care that might be dictated by sound clinical judgement.

The choice of antibiotics will vary between center and will be the antibiotic regimen that is current standard of care in that center. This is due to (i) varying antibiotic regimes among participating centers at present influenced by local factors, including antimicrobial stewardship and drug cost (26) and (ii) a lack of evidence to support a specific antibiotic regimen for childhood appendicitis. Allowing each center to maintain current antibiotic protocols will improve study feasibility and increase generalizability of the results. However, the duration of combined intravenous and oral therapy will be standardized to 10 days.

Following discharge, children who receive non-operative treatment will not be offered elective appendectomy. They will be counselled about the risk of recurrence as part of the permission process for the trial using best available current data. Recurrence of appendicitis within the 1 year follow-up period will be treated with appendectomy; these children will not be eligible for re-enrollment.

Appendectomy group: Children allocated to appendectomy will undergo laparoscopic appendectomy within approximately 18 hours of randomization which is the current standard of care in all centers participating in this study. Participants will receive intravenous antibiotics from the time of randomization and be treated post-operatively with intravenous antibiotics according to a defined and standardized treatment regime based on consensus for this trial. Specifically, children with a macroscopically normal appendix or non-perforated acute appendicitis will receive no further antibiotics. Children with perforated appendicitis will continue to receive intravenous antibiotics for a minimum of 3 days, and may receive additional antibiotics per local practice. The type of antibiotics used in each center will be identical to those used in the non-operative treatment group. Following cessation of intravenous antibiotics, criteria for discharge home will be identical to those in the non-operative treatment group.

ELIGIBILITY:
Inclusion criteria

* children (age 5-16 years)
* clinical and /or radiological diagnosis (ultrasound [US] and/or CT scan) of acute non-perforated appendicitis
* written informed parental/legal guardian permission in accordance with local regulations and institutional policy
* written informed child assent or waiver in accordance with local regulations and institutional policy

Exclusion criteria

* suspicion of perforated appendicitis
* presentation with an appendix mass or phlegmon (on physical examination and/or imaging)
* non-operative management (2 or more rounds of intravenous antibiotics) initiated at an outside institution
* previous episode of appendicitis or appendix mass/phlegmon treated non-operatively
* current treatment for malignancy
* positive pregnancy test (if part of a clinical routine)
* diagnosis of Cystic Fibrosis (CF)

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 978 (Actual)
Dates: Start 2016-01-20; Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
treatment failure | within 1 year of randomization
  The primary outcome is treatment failure. Treatment failure is defined as: (i) additional intervention related to appendicitis requiring general anesthesia within 1 year of randomization (this includes the recurrence of appendicitis after non-operative treatment, which will be treated with appendectomy) or (ii) negative appendectomy. This definition of the primary outcome will capture all important parameters in both treatment groups including specifically: failure of antibiotic treatment requiring appendectomy, significant complication (defined as requiring general anaesthesia) in either treatment group, recurrence of acute appendicitis (treated by appendectomy) and negative appendectomy.

SECONDARY OUTCOMES:
treatment efficacy | within 1 year of randomization
  Secondary outcomes are objective measures of treatment efficacy that fulfil important core areas of relevance to clinicians and patients (pathophysiological manifestations, life impact, resource use and death)
complications | within 1 year of randomization
  complications: adverse events related to non-operative treatment of appendicitis or appendectomy which require additional interventions without general anesthesia, during the first year following randomization
time to discharge | 1 year from randomization
  time to discharge home after randomization measured in hours
number and duration of hospital admissions | within 1 year of randomization
  number and duration of hospital admissions related to appendicitis, appendectomy or their complications during the first year following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Peter SD, Noel-MacDonnell JR, Hall NJ, Eaton S, Suominen JS, Wester T, Svensson JF, Almstrom M, Muenks EP, Beaudin M, Piche N, Brindle M, MacRobie A, Keijzer R, Engstrand Lilja H, Kassa AM, Jancelewicz T, Butter A, Davidson J, Skarsgard E, Te-Lu Y, Nah S, Willan AR, Pierro A. Appendicectomy versus antibiotics for acute uncomplicated appendicitis in children: an open-label, international, multicentre, randomised, non-inferiority trial. Lancet. 2025 Jan 18;405(10474):233-240. doi: 10.1016/S0140-6736(24)02420-6. PMID 39826968
- [Derived] Hall NJ, Eaton S, Abbo O, Arnaud AP, Beaudin M, Brindle M, Butter A, Davies D, Jancelewicz T, Johnson K, Keijzer R, Lapidus-Krol E, Offringa M, Piche N, Rintala R, Skarsgard E, Svensson JF, Ungar WJ, Wester T, Willan AR, Zani A, St Peter SD, Pierro A. Appendectomy versus non-operative treatment for acute uncomplicated appendicitis in children: study protocol for a multicentre, open-label, non-inferiority, randomised controlled trial. BMJ Paediatr Open. 2017 May 18;1(1):bmjpo-2017-000028. doi: 10.1136/bmjpo-2017-000028. eCollection 2017. PMID 29637088